CLINICAL TRIAL: NCT04916860
Title: Clinical Study of SenL-T7 CAR T Cells in the Treatment of Relapsed and Refractory CD7+ T-cell Lymphoblastic Leukemia or T-cell Lymphoblastic Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SenL-T7 for CD7+leukemia/T-LBL
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: SenL-T7 CAR T Cells for CD7+ T-cell Lymphoblastic Leukemia or T-cell Lymphoblastic Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD7 CAR-T (Experimental)
  Interventions: Biological: Senl-T7

INTERVENTIONS:
Biological: Senl-T7 — Patients will be treated with CD7 CAR-T cells

SUMMARY:
This is an open, single-arm, clinical study to evaluate efficacy and safety of anti CD7 CAR-T cell in the treatment of relapsed and refractory CD7+ T-cell lymphoblastic leukemia or T-cell lymphoblastic lymphoma

DETAILED DESCRIPTION:
This study is an open, prospective, dose-increasing clinical study with patients with relapsed or refractory CD7+ T-cell lymphoblastic leukemia or T-cell lymphoblastic lymphoma as subjects. In order to evaluate the safety and efficacy of SENL-T7 in patients with CD7+ T-cell lymphoblastic leukemia or T-cell lymphoblastic lymphoma, the PK/PD indicators of SENL-T7 are also collected. In this study, no dose grouping is set, and 0.5-2E6 /kg× actual body weight dose is selected for reinfusion according to patients' disease diagnosis and tumor load.

The Main research objectives:

To evaluate the safety and efficacy of SENL-T7 in patients with relapsed or refractory CD7+ T-cell lymphoblastic leukemia or T-cell lymphoblastic lymphoma.

The Secondary research objectives:

To investigate the cellular dynamics of SENL-T7 CAR T cells in patients with relapsed or refractory CD7+ T-cell lymphoblastic leukemia or T-cell lymphoblastic lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of relapsed/refractory T-cell lymphoblastic leukemia or T-cell lymphoblastic lymphoma: Induction therapy failed to achieve a complete remission of minor residual negative; Recurrence: after complete remission, any tumor load in the peripheral blood or bone marrow was 5%, or slightly residual positive, or new extramedullary lesions occurred；
2. CD7 expression in tumor cells was detected by flow cytometry；
3. Life expectancy greater than 12 weeks；
4. KPS or Lansky score≥60;
5. HGB≥70g/L (can be transfused);
6. 2-70 years old;
7. oxygen saturation of blood#90%#;
8. Total bilirubin (TBil)≤3 × upper limit normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal;
9. Informed consent explained to, understood by and signed by patient/ guardian.

Exclusion Criteria:

1. Any of the following cardiac criteria: Atrial fibrillation/flutter; Myocardial infarction within the last 12 months; Prolonged QT syndrome or secondary prolonged QT, per investigator discretion. Cardiac echocardiography with LVSF (left ventricular shortening fraction)<30% or LVEF(left ventricular ejection fraction)<50%; or clinically significant pericardial effusion. Cardiac dysfunction NYHA(New York Heart Association) III or IV (Confirmation of absence of these conditions on echocardiogram within 12 months of treatment);
2. Has an active GvHD;
3. Has a history of severe pulmonary function damaging;
4. With other tumors which is/are in advanced malignant and has/have systemic metastasis;
5. Severe or persistent infection that cannot be effectively controlled;
6. Merging severe autoimmune diseases or immunodeficiency disease;
7. Patients with active hepatitis B or hepatitis C([HBVDNA+]or [HCVRNA

   +]);
8. Patients with HIV infection or syphilis infection;
9. Has a history of serious allergies on Biological products (including antibiotics);
10. Clinically significant viral infection or uncontrolled viral reactivation of EBV(Epstein-Barr virus), CMV(cytomegalovirus), ADV(adenovirus), BKvirus, or HHV(human herpesvirus)-6.
11. Presence of symptomatic disorders of the central nervous system, which include but not limited to uncontrolled epilepsy, cerebrovascular ischemia/hemorrhage, dementia, and cerebellar disease, etc.;
12. Have received transplant treatment for less than 6 months in prior to enrollment;
13. Being pregnant and lactating or having pregnancy within 12 months;
14. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First 1 month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after CD7 CAR-T infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Remission Rate | 3 months post CAR-T cells infusion
  To obsere the efficacy of CAR-T cells after infusion, complete remission (CR), complete remission with incomplete recovery of blood cells (CRi), minimal tumor residual positive(MRD+) or negative (MRD-) CR/CRi, disease recurrence or progression (PD) will be used for evaluation.

SECONDARY OUTCOMES:
duration of response (DOR) | 24 months post CAR-T cells infusion
  duration of response (DOR)
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of CD7 CAR- T cells in the genomes of PBMC by qPCR method
progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
Cytokine release | First 1 month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry
CAR-T proliferation | 3 months post CAR-T cells infusion
  percentage of CD7 CAR- T cells measured by flow cytometry method

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei yanda Ludaopei Hospital, Beijingcun, Hebei, China